CLINICAL TRIAL: NCT05054244
Title: Biofilm in Chronic Wound - Clinical Implications and Diagnostic Possibilities
Brief Title: Clinical Implications of Biofilm in Chronic Wound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Tanja Batinac, Associate Prof. M.D. PhD., University of Rijeka
Other Study IDs: uniri-pr-biomed-19-7-1488
Record Dates: First submitted 2021-08-16; First posted 2021-09-23 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Wound; Biofilm; Chronic Pain; Quality of Life; Wound Healing
Keywords: Wound; Biofilm; Chronic pain; Quality of Life; Wound Healing; Hyperbaric oxygenation
MeSH Terms: conditions — Wounds and Injuries; Chronic Pain | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: The patients in control group will be evaluated upon enrolment, after 2, 4, 6 weeks, 3, 6, 9, and 12 months, to evaluate the wound characteristics, clinical healing rate and indicators of biofilm and/or infection. The patients will be treated with standard treatment (dressings, debridement, antibiotics and infection control). The dressing will be performed according to wound characteristics with change every two days including primary dressing (alginates, hydrofiber dressing, antimicrobial dressing, gelling fiber dressing), with silver if infected, and secondary protective dressing (foam with polyurethane) in wounds with granulation tissue. The patient related outcome measures will be evaluated assessing intensity and pain characteristics, quality of life, depression, and anxiety by means of standardized questionnaires: visual analogue scale, McGill Pain questionnaire, Wound Quality of Life Index, Health Quality of Life Questionnaire, Beck depression and Beck anxiety inventory.
  Interventions: Other: standard wound treatment
- HBOT group: The patients in HBOT group will be evaluated upon enrolment, after 2, 4, 6 weeks, 3, 6, 9, and 12 months, to evaluate the wound characteristics, clinical healing rate and indicators of biofilm and/or infection. The patients will be treated with standard treatment (dressings, debridement, antibiotics and infection control). The dressing will be performed according to wound characteristics with change every two days including primary dressing (alginates, hydrofiber dressing, antimicrobial dressing, gelling fiber dressing), with silver if infected, and secondary protective dressing (foam with polyurethane) in wounds with granulation tissue.
  The HBOT sessions will be performed 5 days a week in multi-place chamber at 2.4 atm absolute (ATA) and 100% O2. The patient related outcome measures will be evaluated assessing intensity and pain characteristics, quality of life, depression, and anxiety by means of standardized questionnaires as in control group.
  Interventions: Other: standard wound treatment; Procedure: Hyperbaric oxygenation (HBOT)

INTERVENTIONS:
Other: standard wound treatment — Standard treatment includes dressings, debridement, antibiotics, and bacterial load relief. The dressing will be performed according to wound characteristics with change every two days including primary dressing (alginates, hydrofiber dressing, antimicrobial dressing, gelling fiber dressing), with silver if infected, and secondary protective dressing (foam with polyurethane) in wounds with formed granulation tissue. The progression of the wound and the need for specific treatment will be evaluated weekly by dermatologist and vascular surgeon specializing in wound care, and appropriate treatment conducted according to wound assessment (antibiotics, bandage, dressing change, debridement, amputations).
Procedure: Hyperbaric oxygenation (HBOT) — The HBOT sessions will be performed 5 days a week, in multi-place chamber at 2.4 atm absolute (ATA) and 100% O2 with effective treatment lasting for 90 min. The sessions will be supervised by doctors trained in hyperbaric medicine.
  Groups: HBOT group

SUMMARY:
Chronic wounds are important economic and health-care problem. Biofilm has been recognized as a major factor in wound chronicity, delayed healing, and persistent infections, increasing the need for frequent dressing changes, painful debridement and systemic antimicrobial treatments influencing quality of life. In the presence of "un-cultivating" bacteria and limitations of clinical indicators of biofilm presence, there is a need for simple "screening" diagnostic method for biofilm detection. Chronic wounds of different etiology often associated with chronic pain reduce working abilities and cause restrictions in everyday living diminishing patient's quality of life. Efficacy of hyperbaric oxygenation therapy (HBOT) in treating chronic wound and associated infection has been suggested. This observational prospective cohort study will be conducted at the Department of undersea and hyperbaric medicine and Department of dermatovenereology, Clinical Hospital Center Rijeka during 3-year period from 2021. to 2024. including all patients treated due to chronic wound irrespective of the ethology. The patients will be evaluated upon enrolment, after 2, 4, 6 weeks, and 3, 6, 9, 12 months period, to clinically evaluate the wound characteristics, evaluate clinical healing rate, clinical indicators of biofilm and/or infection, need for additional diagnostic or treatment procedures. The patients in both groups (control and HBOT group) will be treated with standard treatment (dressings, debridement, antibiotics, infection control), in addition HBOT sessions will be performed (HBOT group). Impact of chronic wound and both treatment options to patient related outcome measures will be evaluated assessing intensity and pain characteristics, quality of life, depression, and anxiety by means of standardized questionnaires (visual analogue scale, McGill Pain questionnaire, Wound Quality of Life Index, Health Quality of Life Questionnaire, Beck depression and anxiety inventory). Microbiological analyses of swabs/biopsies will be evaluated to determine microbial profile and resistance. Detection and objectivization of biofilm will be evaluated by standard methods on microbiological isolates (Congo red agar, tube method, tissue culture plate method) and confocal scanning laser microscopy, and on clinical samples by light microscopy. Primary and secondary objective will be assessed after 1 year follow-up.

DETAILED DESCRIPTION:
Observational prospective clinical study will be conducted at the Department of undersea and hyperbaric medicine and Department of Dermatovenereology, Clinical Hospital Center Rijeka, Rijeka, Croatia during the 3-year period, from 2021. to 2024. The study will include all patients treated due to chronic wound irrespective of the wound ethology (arterial, diabetic, venous, decubital, combined etiology, posttraumatic, postamputation, burn, and other), 18 years of age and older, that signed informed consent. The patients will be treated with standard methods, i.e., dressings, debridement, antibiotics, and bacterial load relief (control group) and another group will be additionally treated with HBOT (HBOT group). Exclusion criteria of the study is failure to meet one of the inclusion criteria. The patients with contraindications for HBOT, absolute or relative, patients on bleomycin chemotherapy, with chronic obstructive pulmonary disease, previous spontaneous pneumothorax, chronic otitis media or chronic sinusitis, unstable angina pectoris, severe heart failure, severe dementia, history of seizures, claustrophobia, or significant macroangiopathy with absent both distal pulses and no positive response following oxygen provocation test on transcutaneous oximetry that will not benefit from HBOT.

The sample size has been calculated based on the available formula for comparing two independent groups according to qualitative variables with 95% confidence interval. Total sample size in both groups was estimated to be 62 patients (124 patients in total) with expected average of 10-15% patients to drop-out from the study, so calculated total sample size in both groups was estimated to be 70 patients (140 patients in total). Wound healing rate of 90% and higher is expected to be achieved in HBOT group, while expected healing rate in control group is expected to be at least 20% lower after 1 year follow-up. Correspondingly, the same differences are expected to be achieved in control and HBOT group as regarding manifestations of clinical indications of biofilm presence, clinical and laboratory signs of infections.

The patients will be enrolled in the study following eligibility screen, informed consent, collection of patients history and demographic data (age, gender, marital status, children, education level, profession, employment) with special emphasizes to comorbidities and risk factors (diabetes mellitus, obesity, hypertension, cardiovascular diseases, peripheral arterial diseases) physical examination, clinical wound assessment and evaluation including following: wound number; wound location; wound size (width, length and depth in cm, and calculated wound surface in cm2 and wound volume in cm3); wound duration (days); type of the wound (arterial, diabetic, venous, decubital, combined etiology, other); wound status (stagnant, deteriorating, improving, healed); clinical signs of wound infection (heat/warmth, erythema, increased exudate, purulent exudate, increased pain, discolored granulation tissue, friable granulation tissue, oedema, wound foul odour, delayed healing, suspected biofilm; clinical indications of wound biofilm presence (excessive moisture and wound exudate, low-level of erythema, low-level of chronic inflammation, history of antibiotic failure even with appropriate antibiotic or antimicrobial treatment, cycles of recurrent infection/exacerbation, delayed healing, recalcitrant wound to antimicrobial or antibiotic treatment); wound bed status (approximate % of tissues present in the wound bed rated as necrotic, sloughy, granulation, suspected biofilm, epithelialization); exudate level (level, type); condition of surrounding skin (healthy, macerated, dry/eczematous); photo-documentation upon enrolment and at every follow-up according to the protocol. Additional diagnostic procedures will be performed to assess vascular status of the patient and identify the underlying pathophysiology of the wound and the wound type (pulse palpation, Ankle-brachial Pressure Index, toe pressure and radiological imaging, including duplex Doppler ultrasound, magnetic resonance imaging (MRI) and computed tomography (CT) imaging, transcutaneous oximetry), as well as laboratory examination, swabs/biopsies for microbiological examination. Upon enrollment, routine laboratory work-up (C-reactive protein, complete and differentiate blood count, serum interleukin-6 and pro-calcitonin level, fasting blood glucose, glycosylated hemoglobin, kidney, and liver tests) and wound swabs/biopsy for microbiological analyses will be performed, and repeated as indicated during follow-up period due to clinically suspected signs of infection.

The patients in control groups will be evaluated upon enrolment, after 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months period, and in HBOT group after 10, 20, 30 treatments, 3 months, 6 months, 9 months, 12 months, for clinical wound assessment and evaluation, and to evaluate the wound healing rate and status, perform wound assessment, record clinical indications of biofilm presence and/or signs of infection, laboratory findings, wound characteristics, the need for antibiotic treatment and hospitalization and perform photo-documentation.

The patients in both groups will be treated routinely with standard treatment (dressings, debridement, antibiotics, and bacterial load relief). The dressing will be performed according to wound characteristics with change every two days including primary dressing (alginates, hydrofiber dressing, antimicrobial dressing, gelling fiber dressing), with silver if infected, and secondary protective dressing (foam with polyurethane) in wounds with formed granulation tissue. The progression of the wound and the need for specific treatment will be evaluated and recorded weekly by dermatologist and vascular surgeon specializing in wound care, and appropriate treatment conducted according to wound assessment (antibiotics, bandage, dressing change, debridement, amputations).

In HBOT group, in addition to standard treatment, the HBOT sessions will be performed 5 days a week, in multi-place chamber at 2.4 atm absolute (ATA) and 100% O2 with effective treatment lasting for 90 min. The sessions will be supervised by doctors trained in hyperbaric medicine.

Impact of chronic wound and both, standard and combined treatment, to patient related outcome measures will be evaluated assessing intensity and pain characteristics, quality of life, depression, and anxiety by means of standardized questionnaires. Intensity and characteristics of pain will be evaluated using self-assessment scales for evaluating pain: visual analogue scale -VAS (measured while dressings are in situ, at dressing change, during debridement, 30 min after dressing change or debridement), and McGill Pain questionnaire upon enrolment, after 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months period. Questionaries for evaluating quality of life and overall health state of patient will be performed upon enrolment, after 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months period including: Wound Quality of Life Index (Wound-QoL) and Health Quality of Life Questionnaire (EQ-5D), and questionaries for evaluating depression and anxiety (Beck depression inventory, Beck anxiety inventory) will be performed upon enrolment, after 6 weeks, 3 months, 6 months, 9 months, 12 months period.

Additionally, microbiological analyses of swabs/biopsies will be evaluated using standardized, routine microbiological, cultural, and automatized procedures, to determine microbial profile, differences, and microbial resistance. In addition, detection and objectivization of biofilm will be evaluated using standard methods for biofilm detection (Tissue culture plate method, Congo red agar method, Tube method), confocal scanning laser microscopy (using FilmTracer LIVE/DEAD fluorescence assay and FilmTracer SYPRO Ruby Biofilm Matrix stain, Invitrogen), and on clinical samples, by light microscopy and different staining methods and procedures (Gram stain, Giemsa stain, Crystal violet stain, Congo red stain, Periodic acid-Schiff stain, Hematoxylin and eosin stain).

ELIGIBILITY:
Inclusion Criteria:

* all patients with chronic wound
* chronic wound irrespective of the ethology (arterial, diabetic, venous, decubital, combined etiology, posttraumatic, postamputation, burn, and other)
* 18 years of age and older
* signed informed consent

Exclusion criteria:

• failure to meet one of the inclusion criteria

Exclusion criteria from HBOT group:

* patients with absolute or relative contraindications for HBOT
* patients on bleomycin chemotherapy
* patients with chronic obstructive pulmonary disease, previous spontaneous pneumothorax, chronic otitis media or chronic sinusitis, unstable angina pectoris, severe heart failure, severe dementia, history of seizures, claustrophobia
* patients with significant macroangiopathy and absent both distal pulses and no positive response following oxygen provocation test on transcutaneous oximetry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated due to chronic wound at Department of undersea and hyperbaric medicine and Department of dermatovenereology, Clinical Hospital Center Rijeka during 3-year period from 2021. to 2024., irrespective of wound ethology, 18 years of age and older. The patients will be treated with standard methods (Control group) and with standard methods+ HBOT (HBOT group).
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
wound healing | 1 year of patient follow up
  In participants of both, control and HBOT group, changes in wound healing from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months will be reported by calculating changes in wound sizes from baseline and evaluation times, based on measured wound width, length, and depth (in cm), measured manually and by high-resolution calibrated digital photographs, and calculated wound surface (expressed in cm2) and wound volume (expressed in cm3). In case of multiple wounds all wounds will be measured. The sizes will be averaged at baseline and at every wound assessment to follow wound progress differences in wound healing or/expanding between baseline and 12-month period will be expressed as binary result. The data at baseline and during follow-up period in both patient groups will be compared.
wound status | 1 year follow up
  Changes in wound status from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months will be reported in participants of both, control and HBOT group will be recorded in four categories: stagnant, deteriorating, improving, healed. Complete wound healing will be defined by complete epithelization. The number of patients in both groups will be expressed as binary result in all four categories during the follow-up period. The data at baseline and during follow-up period in both patient groups will be compared.
clinical signs of wound infection | 1 year follow up
  Changes in clinical signs of wound infection from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months in participants of both, control and HBOT group, will be recorded, evaluated as present or absent (yes/no) as follows: heat/warmth, erythema, increased exudate, purulent exudate, increased pain, discolored granulation tissue, friable granulation tissue, oedema, wound foul odour, delayed healing, suspected biofilm. The number of patients in both groups will be expressed as binary result in all categories during follow-up period. The data at baseline and during follow-up period in both patient groups will be compared.
clinical indications of biofilm presence | 1 year follow up
  Changes in clinical indications of wound biofilm presence during routine clinical wound assessment, from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months in participants of both, control and HBOT group, will be recorded as present or absent (yes/no) as follows: excessive moisture and wound exudate, signs of local infection (low-level of erythema, low-level of chronic inflammation), history of antibiotic failure even with appropriate antibiotic or antimicrobial treatment, cycles of recurrent infection/ exacerbation, delayed healing, recalcitrant wound to antimicrobial or antibiotic treatment. The number of patients in both groups will be expressed as binary result in all categories during the follow-up period. The data at baseline and during follow-up period in both patient groups will be compared.
laboratory signs of infections | 1 year follow up
  In participants of both groups, control and HBOT group, changes in laboratory findings of infection as evaluated by concentrations of serum C reactive protein, interleukin-6 and pro-calcitonin, and the number of leukocytes and neutrophiles in peripheral blood from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months, will be recorded. The values of laboratory findings within reference interval will be rated as negative and increased values as positive. The number of patients in both groups will be expressed as binary result in all categories during the follow-up period. The data at baseline and during follow-up period in both patient groups will be compared.
patient related outcome - pain scores in patients with chronic wounds | 1 year follow up
  In participants of both groups, control and HBOT group, changes in pain scores from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months will be reported on Visual Analogue Scale (VAS). Pain scores will be measured while dressings are in situ, at dressing change, during debridement, 30 min after dressing change or debridement, on scale from 0 representing no pain, to 10, latter corresponding to the worst pain and outcome, and expressed as binary result. The data from questionnaire at baseline and during follow-up period in both patient groups will be compared.
patient related outcome - pain quality and intensity in patients with chronic wounds | 1 year follow up
  In participants of both groups, control and HBOT group, changes in sensory and affective pain quality and intensity from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months will be measured by means of standardized McGill Pain questionnaire using 4-point Likert-type scale ranging from 0 to 3. The total score ranges from 0 to 45, latter corresponding to the worse outcome. The data from questionnaire at baseline and during follow-up period in both patient groups will be compared.
patient related outcome - unique overall health state in patients with chronic wounds | 1 year follow up
  In participants of both groups, control and HBOT group, changes in overall patient's health state from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months will be measured by means of standardized questionnaire using Health Quality of Life Questionnaire (EQ-5D), a descriptive system consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), and each dimension has five response levels: 1-no problems, 2-slight problems, 3-moderate problems, 4-severe problems, 5-unable to/extreme problems. A patient's health state is defined by combining one level from each of the five dimensions in a 5-digit code. The data from questionnaire at baseline and during follow-up period in both patient groups will be compared.
patient related outcome - quality of life in patients with chronic wounds | 1 year follow up
  In participants of both groups, control and HBOT group, changes in quality of life from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months will be measured by means of standardized questionnaire using the disease-specific, health-related quality of life of patients with chronic wounds, Wound Quality of Life Index Questionnaire (Wound-QoL) that consists of 17 items on impairments assessed in retrospect to the preceding seven days , and scored with 0 to 4 (0='not at all' to 4='very much'). A Wound-QoL global score on overall disease-specific quality of life will be evaluated computed by averaging all items, with minimal score 0 and highest 68, latter corresponding to the worst outcome. The data from questionnaire at baseline and during follow-up period in both patient groups will be compared.

SECONDARY OUTCOMES:
patient related outcome -depression in patients with chronic wounds | 1 year follow up
  In participants of both groups, control and HBOT group, changes in depression level from baseline and at 6 weeks, 3 months, 6 months, 9 months, 12 months will be performed by means of standardized, self-reported questionnaire, Beck depression inventory with 21-items on a 4-point Likert scale from 0 to 3. The total score ranges from 0 to 63 corresponding to worst outcome. The level of depression is ranged as follows: scores from 1-10 are considered normal, 11-16 - mild mood disturbance, 17-20 borderline clinical depression, 21-30 moderate depression, 31-40 severe depression, and over 40 considered extreme depression and the worst outcome. The data from questionnaire at baseline and during follow-up period in both patient groups will be compared.
patient related outcome - anxiety in patients with chronic wounds | 1 year follow up
  In participants of both groups, control and HBOT group, changes in anxiety level from baseline and at 6 weeks, 3 months, 6 months, 9 months, 12 months will be performed by means of standardized, self-reported questionnaire, Beck anxiety inventory with 21 items on a 4-point Likert scale from 0 to 3. The total score ranges from 0 to 63 corresponding to the worst outcome. The level of anxiety is ranged as follows: scores from 0-7 considered minimal anxiety, 8-15 -mild anxiety, 16-25 - moderate anxiety, and scores 26-63 are considered severe anxiety and the worst outcome. The data from questionnaire at baseline and during follow-up period in both patient groups will be compared.
objectivization of biofilm | 3 years
  Changes in biofilm objectivization from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months will be recorded in participants of both, control and HBOT group, as assessed by standard methods for biofilm detection (Tissue culture plate method, Congo red agar method, Tube method), and confocal scanning laser microscopy (using FilmTracer LIVE/DEAD fluorescence assay and FilmTracer SYPRO Ruby Biofilm Matrix stain, Invitrogen), evaluated as positive and negative. The number of positive/negative samples in both groups will be expressed as binary result for all methods. The data at baseline and during follow-up period in both patient groups will be compared.
clinical screening for the presence of biofilm by light microscopy | 3 years
  Changes in clinical screening for the presence of biofilm from baseline and at 2, 4, 6 weeks, 3 months, 6 months, 9 months, 12 months in participants of both, control and HBOT group, will be recorded, as assessed by light microscopy and different staining methods and procedures on clinical samples (Gram stain, Giemsa stain, Crystal violet stain, Congo red stain, Periodic acid-Schiff stain, Hematoxylin and eosin stain), to evaluate the presence of the following criteria: microbial surface attachment, microbial cells aggregates and exopolymer matrix, will be recorded. The results will be rated as positive in case of two and more criteria present and negative in case of only one. The number of positive/negative samples in both groups will be expressed as binary result. The data at baseline and during follow-up period and data obtained by standard methods for biofilm detection in both patient groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Batinac, M.D., PhD., Principal Investigator — Department of undersea and hyperbaric medicine
Locations (1):
- Department of undersea and hyperbaric medicine, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No